CLINICAL TRIAL: NCT04162379
Title: Effect of Salutatory Oral Prednisolone Dosing on Cancer Pain WHO Stepladder Analgesic Drug Protocol
Brief Title: Oral Prednisolone Effect on Cancer WHO Stepladder Analgesia Protocol
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mohamed Abd Latif Ghanim, Associate Professor os anesthesia ICU & Pain medicine., Mansoura University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R.19.10.656.R1
Record Dates: First submitted 2019-11-11; First posted 2019-11-14 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Steroid Anlgesia in Cancer Pain
Keywords: Steroid, analgesia, Prednisolone, Cancer, cancer Pain, pain WHO stepladder.
MeSH Terms: conditions — Agnosia; Neoplasms; Cancer Pain | interventions — Tablets

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prospective quizi-pre-post oral predensolone (Other): single group and will take oral prednisolone (sulopride10 mg) single dose every two days for 4 successive weeks then the next two weeks as washout period (stop dosing gradually by taking 5 mgs for 3 successive dosing every 2nd day over a week, then stop the oral steroid drug totally over the 2nd week of the washout period. The second period of the study will start by taking the oral prednisolone (sulopride10 mg) every fourth day for the next 4 weeks after which the patient will get another washout two weeks period (stop dosing gradually 5 mgs for 3 successive dosing every 4th day then stop the drug totally).
  Interventions: Drug: Oral tablet

INTERVENTIONS:
Drug: Oral tablet — Patients will be allocated as single group and will take oral prednisolone (sulopride10 mg) single dose every two days for 4 successive weeks then the next two weeks as washout period (stop dosing gradually by taking 5 mgs for 3 successive dosing every 2nd day over a week, then stop the oral steroid drug totally over the 2nd week of the washout period. The second period of the study will start by taking the oral prednisolone (sulopride10 mg) every fourth day for the next 4 weeks after which the patient will get another washout two weeks period (stop dosing gradually 5 mg for 3 successive dosing every 4th day then stop the drug totally).
  Other Names: oral adjuvant analgesia

SUMMARY:
Introduction; World Health Organization (WHO) analgesic ladder; Step I recommends non-opioid analgesics for mild pain. Step II specifies the use of weak opioids for moderate pain. Step III comprises the use of strong opioids for severe pain. Cancer pain management using opioids administered alone or in combination with adjuvant analgesics. Corticosteroids adjuvant use for neuropathic and bone pain treatment. However, despite widespread use of corticosteroids, scientific evidence about its efficacy in cancer pain management is limited. This protocol aims to clarify pors and cons of interrupted steroid dosing in chronic cancer pain WHO stepladder analgesia protocol. Methods; Prospective quizi-pre-post experimental study will be conducted after IRB approval in the Mansoura oncology canter pain clinic-Faculty of medicine Mansoura University Egypt. Verbal informed consent will be obtained from the respondents (patients) for the interview. Furthermore, the data collected from each patient will be kept confidential and used strictly only for the purpose of the study.

Patients will be allocated as single group and will take oral prednisolone (sulopride10 mg) single dose every two days for 4 successive weeks then the next two weeks as washout period (stop dosing gradually by taking 5 mgs for 3 successive dosing every 2nd day over a week, then stop the oral steroid drug totally over the 2nd week of the washout period. The second period of the study will start by taking the oral prednisolone (sulopride10 mg) every fourth day for the next 4 weeks after which the patient will get another washout two weeks period (stop dosing gradually 5 mgs for 3 successive dosing every 4th day then stop the drug totally).A questionnaire-based interview using Brief Pain Inventory-Short Form (BPI-sf) (16) based on VAS pain score as a rough tool for pain intensity Data collection: Primary Outcome: global Pain intensity, assessed by a visual analogue scale (VAS) 0-10. Secondary outcomes based on the Brief Pain Inventory short form (BPI-sf).

DETAILED DESCRIPTION:
Introduction: pain in cancer patients is based on the concept of the World Health Organization (WHO) analgesic ladder and was recently updated with the EAPC (European Association for Palliative Care) recommendations. (1) Cancer pain management using opioids administered alone or in combination with adjuvant analgesics. Spinal cord compression, superior vena cava obstruction, raised intracranial pressure, and bowel obstruction is better established than in other nonspecific indications Corticosteroids adjuvant use for neuropathic and bone pain treatment. However, despite widespread use of corticosteroids, scientific evidence about its efficacy in cancer pain management is limited. According to the cancer Pain Management Index (PMI) (2), approximately one-third of patients do not receive appropriate analgesia proportional to their pain intensity (PI). This protocol aims to clarify pors and cons of interrupted steroid dosing in chronic cancer pain WHO stepladder analgesia protocol.

World Health Organization (WHO) analgesic ladder; Step I recommends non-opioid analgesics for mild pain. Step II specifies the use of weak opioids for moderate pain. Step III comprises the use of strong opioids for severe pain (4). Recently the European Association for Palliative Care (EAPC) recommendations (5, 6). Nociceptive and neuropathic components of cancer pain responsiveness to opioids is necessary to achieve good pain alleviation. Medical data demonstrate that complete pain relief is rarely achieved in cancer patients; nonetheless, it can be significantly reduced (7). However, some authors have suggested eliminating the second step of the analgesic ladder, with weak opioids being replaced with low doses of oral morphine (8, 9).

Inadequate assessment leads to inadequate management of cancer pain. Brief Pain Inventory (PI), a pain assessment tool that measures both the intensity of the pain (sensory dimension) and the interference of cancer pain in the patient's life (reactive dimension). It also queries the patient about pain relief, pain quality, and patient perception of the cause of pain. (10) The Pain Management Index (PMI) is widely used in the assessment of pain management, and negative scores are traditionally considered to indicate inadequate pain management. PMI scores are inversely associated with the proportion of patients with pain interference (PI). However, PMI scores of - 1 do not always indicate inadequate pain management; pain management should, therefore, be evaluated from multiple perspectives.

Hypothalamic-pituitary-Adrenal Axis (HPA) axis, sudden cessation of corticosteroid therapy may result in adrenal failure. Clinically significant HPA axis suppression is rare if a steroid is administered for less than 3 weeks (11). Steroid withdrawal syndromes: Relapse of the disease, symptoms of steroid withdrawal syndrome such as lethargy, depression, anorexia, nausea, myalgia, or arthralgia (12). Steroid Tapering: The most suitable method of tapering has not been established as yet. After the glucocorticoid withdrawal, the hypothalamic and pituitary functions recover first, followed by the adrenocortical function. Full recovery of adrenal function can take months, or even up to a year (13), especially after prolonged steroid treatment with high doses. A possible scheme of steroid discontinuation is Prednisolone or equivalent daily dose≥ 7.5 mg reduce rapidly 2.5 mg every 3-4 days, then 5-7.5 mg reduce by 1 mg every 2-4 weeks, then < 5 mg Reduce by 1 mg every 2-4 weeks (13).

Prednisolone relative biologic potencies are; Salt retention 0.75, Anti-inflammatory effect 3, and HPA axis suppression 4. Nociception consists of four stages: Transduction (in peripheral nociceptors), transmission (via neurons), modulation, and pain perception. The possible role of steroids on every step of remain unclear; Reduction in inflammation decreases nociceptors activation (14) , inhibit the expression of collagenase, reduce pro-inflammatory cytokines, stimulate the synthesis of lipocortin (15), reduction of peritumoral edema leads to the improvement in analgesia in brain metastases (16) and spinal cord compression (17) , Decrease of spontaneous discharge & reduce neuropathic pain, Modulate neural activity and plasticity. There has been little evidence for this in the literature with cancer-induced pain, nausea, and vomiting, fatigue, cancer-induced anorexia-cachexia, depressed mood, or poor general well-being and dyspnea. (18)

ELIGIBILITY:
Inclusion Criteria: Patients will be considered eligible if they fulfill the following criteria: age≥ 18 years old; diagnosed with any type of cancer: on regular visits every 14 days to the Mansoura oncology center pain clinic.

Exclusion Criteria:

patients with severe other medical disease (organ failure-uncontrolled DM-uncontrolled Hypertension) or psychiatric problems and unable or unwilling to provide the required information will be excluded from the study, patients on chemotherapy or radiotherapy during the study period.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Pain intensity: visual analogue scale | from day one to day 28
  global Pain intensity, assessed by a visual analogue scale (VAS) 0-10.

CONTACTS AND LOCATIONS:
Overall Officials: mohamed Ghanem, A professor, Principal Investigator — Mansoura Univeristy
Locations (1):
- Oncolgy Center, Mansoura University,, Al Mansurah, Dakahlia Governorate, Egypt